CLINICAL TRIAL: NCT00747552
Title: Intra-Abdominal Hypertension in Neonatal Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Donald Null M.D., University of Utah
Other Study IDs: 13833
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Intra-Abdominal Hypertension
Keywords: IAP measurements; Abdominal compartment syndrome; NICU patients; Intra-abdominal Hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The observational study is designed to determine the feasibility of performing Intra-Abdominal Pressure (IAP) via bladder pressure measurements and of tracking IAP in neonates who require bladder catheterization. Correlation of IAP measurements with clinical status of the neonatal abdomen will help determine threshold values for Intra-Abdominal Hypertension (IAH) in the neonate.

DETAILED DESCRIPTION:
An increasingly common cause of Multiple Organ Dysfunction Syndrome (MODS) is mechanical injury/ischemia caused by elevated pressures within the abdominal cavity. This phenomenon has been termed intra-abdominal hypertension (IAH) with the final pathway of multiple organ dysfunction and failure termed abdominal compartment syndrome (ACS). In the neonate, IAH is known to accompany omphalocele, gastroschisis and diaphragmatic hernia repair. IAH has also been found to cause a need for neonatal extra corporeal membrane oxygenation (ECMO) and/or a subsequent failure of ECMO treatment.

While abdominal compartment syndrome is the final physiologic and clinically apparent expression of severe elevations of intra-abdominal pressure, earlier in the course of this process, significant organ dysfunction occurs at a sub-clinical level. If mild to moderately elevated abdominal pressure can be detected early, it may allow clinicians to intervene early and reverse the process, preventing progression to ACS and possibly reducing morbidity and mortality.

To date no study has investigated the correlation between bladder pressure (a surrogate measure of IAP) in neonates who may or may not have ACS. Thus, the ranges of normal and elevated IAP are not determined. There is suggestion from pediatric ICU patients that the threshold for IAH in children is less than that in adults. Likewise, the threshold for IAH in neonates may be expected to be even lower, but this remains to be determined.

In this study, IAP (via bladder pressure measurements) will be measured with a commercially available and FDA approved system which utilizes an electronic pressure transducer, tubing, and any bedside patient monitor with pressure measurement inputs. These types of monitors are standard in the NICU. The pressure transducer is attached to the bladder catheter via a two-way valve, allowing urine drainage in-between taking bladder pressure measurements. A small amount of sterile saline is infused into the bladder in order to make the IAP measurement. While there is an indwelling urinary catheter, bladder pressure measurements will be taken every 2-4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Any NICU patient is eligible for enrollment in this study if his/her medical condition has required the placement of a bladder catheter for urine drainage and who does not meet any of the following Exclusion Criteria.

Exclusion Criteria:

* Bladder trauma
* History of recent bladder surgery
* Neurogenic bladder

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective observational study. A convenience sample of 50 NICU patients will be planned to be enrolled at Primary Children's Medical Center and/or the University of Utah Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald .Null, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah / Primary Childrens Medical Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Jan 2006 to Apr 2008, 32 infants who were inpatients in NICU were enrolled into the study.
Pre-assignment Details: 2 of the infants that were enrolled had the urinary catheter removed prior to any data collection. As the presence of a urinary catheter is necessary for bladder measurements, no data was able to be collected and therefore never actually started in the study.
Groups:
- Infants With Urinary Catheter in Place: Any infant admitted to the NICU who requires an indwelling urinary catheter as part of their illness will qualify for this study. This group will be further analyzed based on whether their illness is due to abdominal abnormalities or disease or whether there is another serious illness requiring an indwelling urinary catheter. The group will also be analyzed pre and post-operatively.
Period: Overall Study
Arm/Group | Infants With Urinary Catheter in Place
Started | 30 (This number does not include the 2 who were enrolled but had no data collected on them.)
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infants With Urinary Catheter in Place
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Intra-abdominal Pressure(IAP) Measurements in NICU Patients.
Description: Intra-abdominal Pressure (IAP) measurements were taken using an electronic pressure transducer via an indwelling urinary catheter. Measurements were obtained every 2-4 hours while the urinary catheter remained in place. This will be used to determine feasability of using a urinary catheter and electronic pressure transducer system to determine IAP. A total of 1219 measurements were obtained from 30 subjects.
Time Frame: 3 years
Population: 18 of the neonates required staged abdominal surgery for various abdominal abnormalities or disease, while 12 of the neonates were ill due to PPHN, sepsis, or hydrops. All analysis was per protocol.
Measure: Number; unit: IAP measurements
Arm/Group | Infants With Urinary Catheter in Place
Number analyzed (Participants) | 30
IAP measurements | 1219

2. Secondary Outcome: Median Bladder Pressure for All Measurements
Description: Intra-abdominal Pressure (IAP) measurements will be tabulated and frequency distributions determined for patients with and without any clinical/surgical abdominal pathology. Median and quartile values will be assessed in order to describe normative values. In patients with clinical abdominal pathology (abdominal distention, necrotizing enterocolitis, abdominal wall defects, diaphragmatic hernia, etc), sequential evaluation of IAP will be done to try to identify thresholds for Intra-abdominal Hypertension (IAH).
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Infants With Urinary Catheter in Place
Number analyzed (Participants) | 30
mmHg | 8 (7.1) [3 to 10]

ADVERSE EVENTS:
Arm/Group | Infants With Urinary Catheter in Place
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No